CLINICAL TRIAL: NCT03178877
Title: The Prevalence of Irritable Bowel Syndrome Using Rome IV Criteria in Medical Student and The Related Factors
Acronym: IBS
Status: Completed | Type: Observational
Sponsor: Indonesia University (Other)
Responsible Party: Principal Investigator, Ari Fahrial Syam, Medical Doctor, Gastroenterology Hepatology Consultant, Indonesia University
Other Study IDs: 16-11-430
Record Dates: First submitted 2017-06-03; First posted 2017-06-07 (Actual); Last update posted 2017-06-07 (Actual); Status verified 2017-06

CONDITIONS: IBS - Irritable Bowel Syndrome
Keywords: IBS, Rome IV criteria, anxiety
MeSH Terms: conditions — Irritable Bowel Syndrome; Ichthyosis Bullosa of Siemens; Anxiety Disorders

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- IBS: IBS group is medical student who filled Rome IV criteria for IBS
  Interventions: Other: No intervention
- Non IBS: Non-IBS group is non IBS medical student based on Rome IV criteria
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention

SUMMARY:
A cross-sectional study of 350 medical student Universitas Indonesia from first grade until fifth grade was done during November-December 2016. This study used stratified randomized sampling. The Rome IV criteria was used for diagnosing IBS. Questionnaire-guided interview was applied to all subjects.

DETAILED DESCRIPTION:
A cross-sectional study of 350 medical student Universitas Indonesia from first grade until fifth grade was done during November-December 2016. This study used stratified randomized sampling. The Rome IV criteria was used for diagnosing IBS. Questionnaire-guided interview was applied to all subjects. A bivariate analysis was done to know the relationship between IBS and its related factors using chi-square, unpaired t-test, and their alternatives. Multivariate analysis was done using logistic regression test

ELIGIBILITY:
Inclusion Criteria:

* Age of participant >= 15 years
* Volunteer to participate in study

Exclusion Criteria:

* Red flag symptoms: febrile, vomiting, rectal bleeding, weight lost
* Diagnosed as having Inflammatory bowel disease
* Peptic ulcer drug consumption
* History of gastrointestinal surgery

Ages: 15 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Medical student from first grade to fifth grade
Sampling Method: Probability Sample
Enrollment: 350 (Actual)
Dates: Start 2016-11-01 (Actual); Primary Completion 2016-12-31 (Actual); Study Completion 2016-12-31 (Actual)

PRIMARY OUTCOMES:
Anxiety and depression | 1 month
  Anxiety and Depression using Hospital Anxiety Depression Scale

SECONDARY OUTCOMES:
Sleep Quality | 1 month
  Sleep quality using Pittsburg Sleep Quality Index
Spiritual status | 1 month
  Spiritual status using Functional Assessment of Chronic Illness Therapy-Spiritual Wellbeing
Academic Stress | 6 months
  Academic stress using Student-Life Stress Inventory

CONTACTS AND LOCATIONS:
Locations (1):
- Cipto Mangunkusumo Hospital, Jakarta Pusat, DKI Jakarta, Indonesia

IPD SHARING:
Plan to Share IPD: No
Not available to other researcher